CLINICAL TRIAL: NCT05043402
Title: An Open Label Randomized Study of Navicixizumab Plus Paclitaxel and Navicixizumab Monotherapy in Comparison to Paclitaxel Monotherapy in Patients With Platinum-Resistant Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: A Study of Navicixizumab in Patients With Platinum Resistant Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: OncXerna Theraputics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONCX-NAV-G301; 2021-001933-38 (EudraCT Number)
Record Dates: First submitted 2021-09-07; First posted 2021-09-14 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Platinum-Resistant
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — navicixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Combination navicixizumab + paclitaxel (Experimental): Combination navicixizumab + paclitaxel: navicixizumab 3 mg/kg Q2W of a 28 day cycle (i.e., Days 1 and 15); paclitaxel 80 mg/m2 on Days 1, 8 and 15 of a 28 day cycle
  Interventions: Drug: navicixizumab; Device: Xerna™ TME Panel
- Paclitaxel monotherapy (Active Comparator): Paclitaxel monotherapy: paclitaxel 80 mg/m2 on Days 1, 8 and 15 of a 28-day cycle
  Interventions: Device: Xerna™ TME Panel
- Navicixizumab monotherapy (Experimental): Navicixizumab monotherapy: navicixizumab 3 mg/kg Q2W of a 28-day cycle (i.e., Days 1 and 15)
  Interventions: Drug: navicixizumab; Device: Xerna™ TME Panel

INTERVENTIONS:
Drug: navicixizumab — navicixizumab IV
  Other Names: navi
  Arms: Combination navicixizumab + paclitaxel; Navicixizumab monotherapy
Device: Xerna™ TME Panel — RNA-seq-based biomarker platform that classifies any given patient tumor sample into phenotypes based on the dominant biology of the tumor microenvironment (TME).

SUMMARY:
This is a Phase 3, randomized, open-label, 2-stage, multicenter study of navicixizumab with or without paclitaxel compared with paclitaxel monotherapy in patients with platinum-resistant advanced epithelial ovarian cancer and specific biomarkers, as measured by the proprietary and validated Xerna™ TME Panel biomarker assay. Eligible patients must have received at least 2 prior regimens but not more than 5 prior regimens, including treatment with a monoclonal antibody angiogenesis inhibitor (e.g., bevacizumab), must be considered platinum-resistant, and must be considered appropriate to receive single-agent paclitaxel chemotherapy as a next line of therapy. All patients must be willing and able to provide a formalin-fixed paraffin embedded (FFPE) archive or core tumor sample collected during screening for classification as B+ or B- biomarker status based on RNA expression data from the Xerna™ TME Panel biomarker assay. The co-primary efficacy endpoints are ORR by RECIST v1.1 and PFS (as assessed by blinded independent radiological review [BIRR]) analyzed at different timepoints. Analysis of the ORR primary efficacy endpoints will occur at the end of Stage 1 and at the end of Stage 2; the PFS primary efficacy endpoint will be analyzed at the end of Stage 2.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, open-label, 2-stage, multicenter study of navicixizumab with or without paclitaxel compared with paclitaxel monotherapy in patients with platinum-resistant advanced epithelial ovarian cancer and specific biomarkers, as measured by the proprietary and validated Xerna™ TME Panel biomarker assay. Eligible patients must have received at least 2 prior regimens but not more than 5 prior regimens, including treatment with a monoclonal antibody angiogenesis inhibitor (e.g., bevacizumab), must be considered platinum-resistant, and must be considered appropriate to receive single-agent paclitaxel chemotherapy as a next line of therapy. All patients must be willing and able to provide a formalin-fixed paraffin embedded (FFPE) archive or core tumor sample collected during screening for classification as B+ or B- biomarker status based on RNA expression data from the Xerna™ TME Panel biomarker assay. The co-primary efficacy endpoints are ORR by RECIST v1.1 and PFS (as assessed by blinded independent radiological review [BIRR]) analyzed at different timepoints. Analysis of the ORR primary efficacy endpoints will occur at the end of Stage 1 and at the end of Stage 2; the PFS primary efficacy endpoint will be analyzed at the end of Stage 2.

Patients will be stratified by Xerna™ TME Panel status and region and randomized to the following treatment arms according to the corresponding study stage randomization ratios. Enrollment will proceed from Stage 1 to Stage 2 without interruption:

Stage 1 treatment arms (4:4:1 randomization):

* Combination navicixizumab + paclitaxel: navicixizumab 3 mg/kg once every 2 weeks (Q2W) of a 28-day cycle (i.e., on Days 1 and 15); paclitaxel 80 mg/m2 on Days 1, 8 and 15 of a 28-day cycle
* Paclitaxel monotherapy: paclitaxel 80 mg/m2 on Days 1, 8 and 15 of a 28-day cycle
* Navicixizumab monotherapy: navicixizumab 3 mg/kg Q2W of a 28-day cycle (i.e., on Days 1 and 15)

  • Stage 2 treatment arms (2:2:3 randomization):
* Combination navicixizumab + paclitaxel: navicixizumab 3 mg/kg Q2W of a 28-day cycle (i.e., on Days 1 and 15); paclitaxel 80 mg/m2 on Days 1, 8 and 15 of a 28-day cycle
* Paclitaxel monotherapy: paclitaxel 80 mg/m2 on Days 1, 8 and 15 of a 28-day cycle
* Navicixizumab monotherapy: navicixizumab 3 mg/kg Q2W of a 28-day cycle (i.e., on Days 1 and 15) Within each treatment arm, patients will be stratified to a B+ or B- cohort based on their Xerna™ TME Panel biomarker assay results during screening.

Patients in both stages will have radiologic tumor assessments every 8 weeks (±1 week), regardless of treatment delays, until objective disease progression, initiation of subsequent anticancer therapy, withdrawal of consent, death, or end of study, whichever occurs first. All patients will continue to receive study treatment until progressive disease (PD) per RECIST v1.1 (as assessed by the investigator), the development of unacceptable toxicity, withdrawal of consent, or another protocol-defined discontinuation criteria is met, whichever occurs first, or until the sponsor terminates the study.

Treatment decisions (i.e., whether to continue or discontinue the study medication) should not be made based on CA-125 levels. Progression during protocol treatment cannot be declared on the basis of CA 125 alone.

All patients who discontinue study treatment for any reason will be followed for survival at 3-month intervals until death or withdrawal of consent, whichever occurs first. Survival follow-up will continue for 12 months after the last patient is enrolled or approximately 75% of the population has died, whichever is later.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Patients must have received ≥2 and not more than 5 prior therapies, including at least 1 line of therapy containing bevacizumab (or biosimilar).
* Patients must be considered platinum-resistant, defined as progression within 6 months from completion of a platinum-containing therapy
* Patient must be considered appropriate for treatment with weekly paclitaxel monotherapy as the next line of therapy.
* Patient must be willing and able to provide an FFPE archival or core tumor sample for determination of biomarker status on the Xerna™ TME Panel biomarker assay (positive or negative) prior to study treatment.
* Presence of at least one measurable lesion, as defined by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1 Adequate organ function

Exclusion Criteria:

* Non-epithelial ovarian carcinoma.
* Ovarian tumors with low malignant potential (i.e., borderline tumors).
* Primary platinum-refractory disease (defined as progression during or within 4 weeks after completion of the first platinum regimen).
* Patient has received an anti-angiogenic product other than bevacizumab or biosimilar.
* Patient has congestive heart failure
* Patient has a history of myocardial infarction, cerebral vascular accident, or transient ischemic attacks within 6 months
* Patient has a history of cardiac ischemia or heart failure within 6 months
* Baseline B-type natriuretic peptide (BNP) value >100 pg/mL or N-terminal-proBNP (NT-proBNP) value of > 125 pg/mL.
* LVEF <50%.
* Peak tricuspid velocity >3.0 m/s on Doppler ECHO.
* Clinically significant ECG abnormality, as assessed by the investigator
* Blood pressure (BP) >140/90 mmHg
* History of bowel obstruction, including sub-occlusive disease, related to the underlying disease
* Hemoptysis >2.5 mL within 8 weeks prior
* Major surgical procedure, or significant traumatic injury within 28 days
* Uncontrolled seizure disorder or active neurologic disease
* Patients with a cardiac aneurysm.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 2 years
  Overall Response Rate defined as the proportion of patients with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR), by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
PFS | Up to 2 years
  Progression Free Survival

SECONDARY OUTCOMES:
OS | Up to 2 years
  Overall Survival
TTR | Up to 2 years
  Time to response
DCR | Up to 2 years
  Disease control rate defined as the proportion of patients with stable disease (SD) or a confirmed BOR of CR or PR
DOR | Up to 2 years
  Duration of Response

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen N Moore, MD,MS, Principal Investigator — University of Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961